CLINICAL TRIAL: NCT06889818
Title: Korean Joint Registry for Alzheimer's Treatment and Diagnostics (JOY-ALZ)
Acronym: JOY-ALZ
Status: Recruiting | Type: Observational
Sponsor: Ewha Womans University Mokdong Hospital (Other)
Collaborators: Korean Dementia Association (Unknown); Inha University Hospital (Other); Gachon University Gil Medical Center (Other); Saint Vincent's Hospital, Korea (Other); Gangnam Severance Hospital (Other); Konkuk University Hospital (Other); Kyunghee University Medical Center (Other); Korea University Medicine (Unknown); Busan University Medical Center (Unknown); CHA University (Other); Samsung Medical Center (Other); Seoul National University Hospital (Other); Seoul National University Bundang Hospital (Other); Asan Medical Center (Other); Soonchunhyang University Hospital (Other); Ajou University Hospital, Suwon, South Korea (Unknown); Yonsei University Yongin Severance Hospital (Unknown); Wonkwang University Hospital (Other); Ewha Womans University Seoul Hospital (Other); InjeUniversityBusanPaikHospital (Unknown); Chonnam National University Hospital (Other); Jeju National University Hospital (Other); Chungnam National University Hospital (Other); Gyungbook national university hospital (Unknown); Hanllym University Medical Center (Unknown); Heavenly Clinical Research (Other); KangWon National University Hospital (Other); Seoul St. Mary's Hospital, The Catholic University (Unknown)
Responsible Party: Principal Investigator, Geon Ha Kim, Principal Investigator, Ewha Womans University Mokdong Hospital
Other Study IDs: JOY-ALZ
Record Dates: First submitted 2025-03-14; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-02

CONDITIONS: Mild Cognitive Impairment; Dementia; Subjective Cognitive Decline (SCD); Alzheimer Disease
Keywords: Real World Data; Lecanemab
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Only if agreed, 1.5 tablespoons (23 cc) of blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Open Label Registry: Collection of real-world data from enrolled patients being evaluated for or receiving novel Korea MFDS-approved Alzheimer's disease treatments and diagnostics

SUMMARY:
The purpose of this research is to investigate the long-term effectiveness and safety of new Alzheimer's disease treatments, particularly monoclonal antibody therapies like lecanemab and donanemab, as well as to enhance diagnostic methods for Alzheimer's disease by collecting real-world data from Korean Alzheimer's patients. The goal is to contribute to the precision of Alzheimer's treatment and to evaluate the impact of these new therapies and diagnostic techniques in clinical practice.

DETAILED DESCRIPTION:
In 2024, it is estimated that there will be over 1 million individuals aged 65 and older with dementia in South Korea, with national dementia care costs exceeding approximately 17 trillion KRW (0.9% of GDP). South Korea is experiencing rapid population aging, leading to a projected significant increase in both the number of patients and the associated socio-economic costs. Alzheimer's disease (AD) is the most common cause of dementia and cognitive impairment in the elderly, characterized by the abnormal accumulation of amyloid beta (Aβ) and tau proteins in the brain. Research has shown that beta-amyloid protein begins to accumulate in the brain over 20 years before the onset of memory impairment symptoms. Consequently, Alzheimer's disease progresses through a prolonged asymptomatic stage of normal cognitive function (cognitively unimpaired, CU) to subjective cognitive decline, mild cognitive impairment, and dementia.

In May 2024, the Korean Ministry of Food and Drug Safety approved lecanemab for the treatment of Alzheimer's disease. Recent advancements have been made in the development of new treatments and diagnostic methods for Alzheimer's disease, with some already approved for use in South Korea or anticipated to receive approval soon. These developments are expected to significantly impact the management of dementia and cognitive impairment patients in the near future. Among the new treatments, monoclonal antibody injections targeting the core pathological mechanism of Alzheimer's disease, which is the removal of beta-amyloid protein (e.g., lecanemab, donanemab), currently lack long-term efficacy data, providing only 1-2 years of investigatory data in clinical trials. Such medications may have side effects, including amyloid-related imaging abnormalities (ARIA) such as brain edema or microbleeding and infusion-related adverse reactions. For the advancement of precise treatments for Alzheimer's disease, it is essential to monitor long-term effects and side effects of these drugs in clinical practice to collect and analyze more extensive clinical data to establish additional clinical evidence.

Moreover, the phase 3 clinical trial data for lecanemab suggests that the drug's effectiveness and side effects may vary by ethnicity. Recently, a diagnostic technique that measures Elecsys beta-amyloid 42 (Aβ42) and Elecsys Phospho-Tau181 (ptau181) in cerebrospinal fluid (CSF) has received approval from the Korean Ministry of Food and Drug Safety for the diagnosis of Alzheimer's disease. Additionally, there is a strong potential for new diagnostic methods that measure proteins such as ptau217, ptau181, and Aβ42 in blood to be commercialized in clinical practice. Future advancements through real-world data collection on these new diagnostic methods will be necessary.

The Alzheimer's Association (AA) and researchers in the United States have initiated a registry study named the Alzheimer's Network for Treatment and Diagnostics (ALZ-NET) to collect real-world data on new treatments and diagnostic methods for Alzheimer's disease. Longitudinal studies to investigate the long-term effectiveness and safety of new treatments and diagnostic methods in Alzheimer's patients are also being established in countries such as Japan, Australia, the Netherlands, and Europe. In response to these changes in Alzheimer's disease management, the researchers aim to contribute to the precision of Alzheimer's treatment and the enhancement of new diagnostic methods by collecting real-world data from Korean Alzheimer's patients regarding the long-term effectiveness and safety of new therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be 19 years of age or older at the time of informed consent.
2. Patients who are undergoing medical evaluation for newly approved Alzheimer's disease medications after 2021, patients who have decided to initiate treatment with these medications in consultation with their physician after 2021, or patients who have already started treatment with newly approved Alzheimer's disease medications after 2021.
3. Patients who have undergone an amyloid PET scan to confirm Alzheimer's disease pathology, or cerebrospinal fluid testing for Aβ42 and ptau181.
4. Clinical diagnosis of Alzheimer's disease, defined as follows:

<!-- -->

1. [Alzheimer's Disease Dementia (ADD)] - Must meet the criteria for probable Alzheimer's dementia as defined by the National Institute on Aging and the Alzheimer's Association working groups (NIA-AA).

   * Must exhibit cognitive decline that impairs independent daily living.
2. [Mild Cognitive Impairment (MCI)]

   - Must meet NIA-AA diagnostic criteria for MCI.

   - The subject or informant must report cognitive decline.

   - Performance on delayed recall of verbal memory must be more than -1.0 SD below the age- and education-adjusted normative mean, or scores on any one or more tests of executive function, language, visuospatial abilities, or attention must be more than -1.5 SD below the age- and education-adjusted normative mean.

   - Clinical Dementia Rating scale (CDR) of 0.5.

   - Maintenance of independent daily living ability.

   - Not categorized as dementia.
3. [Cognitively Unimpaired (CU)]

   - Delayed recall of verbal memory must be at or above -1.0 SD versus the age- and education-adjusted normative mean, and all executive function, language, visuospatial abilities, and attention tests must be at or above -1.5 SD versus the age- and education-adjusted normative mean.

   - Maintenance of independent daily living ability.
   * If the subject reports cognitive decline, they will be classified as having Subjective Cognitive Decline (SCD).

     5. Patients must be ambulatory (use of mobility aids is acceptable). 6. The subject must provide written informed consent to participate in the study. In the case of dementia patients, additional written consent from a guardian is required.

Exclusion Criteria:

1. Presence of significant psychiatric disorders associated with intellectual disability, schizophrenia, major depression, bipolar disorder, delirium, etc.
2. History of substance abuse or alcohol dependence that required treatment within the past five years.
3. A current diagnosis of cancer that has not achieved remission within the past five years. However, localized prostate cancer, cervical carcinoma in situ, non-melanoma skin basal cell carcinoma, or squamous cell carcinoma are excluded.
4. Evidence of severe or unstable physical conditions (e.g., dialysis, severe liver disease).
5. Visual or auditory impairments that prevent the satisfactory assessment of cognitive function.
6. Inability to perform MRI due to the presence of metallic substances in the body.
7. Currently participating in another drug clinical trial.
8. Currently pregnant or breastfeeding.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 40 medical institutions nationwide are expected to participate in the study over a period of 10 years, with about 4,000 participants in total. Our institution anticipates the participation of approximately 100 subjects. Participants in this study are adults with Alzheimer's disease dementia, mild cognitive impairment, or normal cognitive function (including subjective cognitive decline) who are undergoing medical evaluation for newly approved Alzheimer's disease medications after 2021, have made the decision to initiate treatment with these medications, or have already begun treatment with these newly approved Alzheimer's disease medications.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2034-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Korean Mini-Mental State Examination-2 (K-MMSE-2) total score | Up to 10 years
  This test consists of orientation to time and place, three-word recall, subtracting 7 from 100 in succession, overlapping pentagon drawing, command execution, reading, writing, repeating, and naming. The score ranges from 0 to 30.
Change from baseline in the Korean version of Montreal Cognitive Assessment (K-MOCA) total score | Up to 10 years
  This assessment evaluates memory, language, executive function, visuospatial construction, reasoning, and attention, with a scoring range of 0-30 points where higher scores indicate better cognitive function.
Change from baseline in the Clinical Dementia Rating scale (CDR) total score | Up to 10 years
  Scores include a Global CDR (0-3 points) and a CDR-Sum of Boxes (SB) which sums the scores of the six domains (0-18 points). Higher scores indicate worse cognitive function.
Change from baseline in the Functional Assessment Questionnaire (FAQ) total score | Up to 10 years
  The informant evaluates the subject, with a score range of 0-30, where higher scores indicate a decline in daily functioning. A score of 9 or more suggests significant deterioration in daily functioning.
Change from baseline in the Korean version of the Alzheimer disease 8 (K-AD8) total score | Up to 10 years
  The score ranges from 0 to 8, where higher scores indicate more severe cognitive impairment.

SECONDARY OUTCOMES:
Brain Magnetic Resonance Imaging (MRI) | Up to 10 years
  Data will be collected to diagnose cognitive impairment and to assess for emergence of amyloid related imaging abnormalities.
Alzheimer's disease (AD) biomarkers | Up to 10 years
  Data from past amyloid Positron Emission Tomography (PET) scans will be collected for the diagnosis of AD. Results for cerebrospinal fluid assays of Elecsys Aβ42, Elecsys ptau181, and ptau181/Aβ42 will also be collected. A ptau181/Aβ42 ratio greater than 0.023 indicates a suggestion of AD.

CONTACTS AND LOCATIONS:
Overall Officials: Geon-ha Kim, Principal Investigator — Ewha Womans University Mokdong Hospital; Seong-hye Choi, Principal Investigator — Inha University Hospital; Kee-hyung Park, Principal Investigator — Gachon University Gil Medical Center
Locations (3):
- South Korea (3):
  - Gachon University Gil medical Center, Incheon
  - Inha University Hospital, Incheon
  - Ewha Womans University Mokdong Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with Eisai and gAAIN.

REFERENCES:
- [Derived] Kim GH, Pyun JM, Kang D, Kang SH, Koh SH, Kim JS, Moon SY, Moon WJ, Park YH, Shim Y, Yang DW, Youn YC, Jung YH, Cho H, Choi H, Lim JS, Park KH, Choi SH. A Protocol of Korean JOint RegistrY for ALZheimer's Treatment and Diagnostics (JOY-ALZ). Dement Neurocogn Disord. 2026 Jan;25(1):25-41. doi: 10.12779/dnd.2026.25.1.25. Epub 2026 Jan 15. PMID 41657474